CLINICAL TRIAL: NCT05518513
Title: Continuous Infusion and Intermittent Bolus Adductor Canal Block for Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Wei-Teng Weng, Attending Physician of Anesthesiology, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCKUH-11109019
Record Dates: First submitted 2022-08-21; First posted 2022-08-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Arthroplasty, Replacement, Knee; Adductor Canal Block
Keywords: total knee arthroplasty; adductor canal block; nerve block; regional analgesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous infusion (Experimental): adductor canal block with continuous infusion of 0.25% bupivacaine 3.5 ml per hour for 2 days postoperatively
  Interventions: Drug: Bupivacain
- 12hrs intermittent bolus (Active Comparator): adductor canal block with intermittent bolus of 0.25% bupivacaine 21 ml every 12 hours for 2 days postoperatively
  Interventions: Drug: Bupivacain
- 6hrs intermittent bolus (Experimental): adductor canal block with intermittent bolus of 0.25% bupivacaine 21 ml every 6 hours for 2 days postoperatively
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — adductor canal block with 0.25% bupivacaine
  Other Names: Marcaine

SUMMARY:
The investigators believed the analgesic efficacy of adductor canal block on patients receiving total knee arthroplasty. However, the analgesic effects of different delivery regimens and duration of effects are variable. The investigators hypothesize that using continuous infusion and shorter interval bolus of local anesthetics to perform adductor canal block will reduce pain scale and opioid consumption in patients receiving total knee arthroplasty compared with longer interval bolus of local anesthetics.

DETAILED DESCRIPTION:
Sensory innervations contributing pain after total knee arthroplasty (TKA) include branches of femoral, obturator and sciatic nerves. Branches of femoral nerve contribute the most pain sensation in TKA including nerves to the vastus medialis, intermedius, and lateralis, medial and intermediate femoral cutaneous, and saphenous nerves. Smaller contribution of pain sensation from branches of fibular and tibial nerves, and posterior branch of obturator nerve. Multiple techniques of nerve block could anesthetize some or all of the sensory innervations, but analgesia with motor sparing is important for early recovery and rehabilitation after TKA. For both pain reduction and motor function, adductor canal block (ACB) combined with local infiltration analgesia is considered more feasible than other peripheral nerve blocks.

ACB could anesthetize nerves beyond in adductor canal. Anatomical studies revealed the extended spreading of local anesthetics (LA) beyond adductor canal when performing ACB, and caudal spreading could reach popliteal fossa through adductor hiatus. Cephalad spreading of LA in ACB is limited and rarely extending to femoral triangle even when injecting from proximal adductor canal, but the cephalad spreading also depends on the volume of injectants and using tourniquets.

In clinical studies, both ACB injection site and volume of injectants were investigated. Clinical trials and systematic reviews revealed the similar efficacy of analgesia when ACB injection at proximal and distal adductor canal, although the volume and pattern of injection (bolus or continuous) were variable. Regarding to the volume of injectants, 20ml injectant of local anesthetics would be adequate without prominent motor impairment compared with smaller volume.

Previous systematic reviews and meta-analysis have confirmed better analgesia with continuous infusion of ACB than single shot, but few studies explored the difference of intermittent bolus and continuous infusion. One clinical trial compared continuous infusion and intermittent bolus of ACB in patients receiving TKA, two other trials investigated the difference in healthy volunteers and patients receiving knee arthroscopy. All these three studies concluded no difference of analgesic efficacy. However, no consistent volume and frequency of injection was studied. Whether longer interval of intermittent bolus was the same with continuous infusion in analgesic efficacy is still need to be further verified.

ELIGIBILITY:
Inclusion Criteria:

* Adults receiving unilateral total knee arthroplasty under spinal anesthesia
* American society of anesthesiologists 1-3

Exclusion Criteria:

* Could not cooperate
* Allergy to medicines used in the study
* Chronic pain
* Long term opioid use
* Neuromuscular disease
* Surgical complication: massive bleeding, postoperative ICU, unanticipated procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Accumulated morphine consumption | In postoperative 48 hours
  Additional morphine prescription

SECONDARY OUTCOMES:
Numerical pain scale at rest | In postoperative 2 days
  From no pain felt as 0 to the most pain felt as 10, measuring pain score at postoperative care unit, 3/9 pm on operative day, 9 am and 3/9 pm on postoperative day 1, 9 am and 3/9 pm on postoperative day 2
Numerical pain scale during knee flexion | In postoperative 2 days
  From no pain felt as 0 to the most pain felt as 10, measuring pain score at postoperative care unit, 3/9 pm on operative day, 9 am and 3/9 pm on postoperative day 1, 9 am and 3/9 pm on postoperative day 2
Percentage of muscle power decrement | In postoperative 2 days
  Extension strength of thigh at surgical side, measurement before surgery and postoperatively, access by dynameter as participants sit and perform surgical leg thigh extension, assessing at 9 am on postoperative day 1 and 2
Postoperative nausea and vomiting | In postoperative 2 days
  Access if any sensation of nausea or episodes of vomiting
Event of falling down | In postoperative 2 days
  Record the number of events of falling down

OTHER OUTCOMES:
Opioid related side effect | In postoperative 2 days
  Record if any sensation of urinary retention, skin pruritus
Nerve block related complication | In postoperative 2 days
  Record if any episode of nerve block insertion site hematoma, leakage of local anesthetics, or local anesthetic systemic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: WEI-TENG WENG, MD, Principal Investigator — Department of Anesthesiology, National Cheng Kung University Hospital, Taiwan
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Result] Monahan AM, Sztain JF, Khatibi B, Furnish TJ, Jaeger P, Sessler DI, Mascha EJ, You J, Wen CH, Nakanote KA, Ilfeld BM. Continuous Adductor Canal Blocks: Does Varying Local Anesthetic Delivery Method (Automatic Repeated Bolus Doses Versus Continuous Basal Infusion) Influence Cutaneous Analgesia and Quadriceps Femoris Strength? A Randomized, Double-Masked, Controlled, Split-Body Volunteer Study. Anesth Analg. 2016 May;122(5):1681-8. doi: 10.1213/ANE.0000000000001182. PMID 26863502
- [Result] Thapa D, Ahuja V, Verma P, Gombar S, Gupta R, Dhiman D. Post-operative analgesia using intermittent vs. continuous adductor canal block technique: a randomized controlled trial. Acta Anaesthesiol Scand. 2016 Nov;60(10):1379-1385. doi: 10.1111/aas.12787. Epub 2016 Sep 4. PMID 27592690
- [Result] Jaeger P, Baggesgaard J, Sorensen JK, Ilfeld BM, Gottschau B, Graungaard B, Dahl JB, Odgaard A, Grevstad U. Adductor Canal Block With Continuous Infusion Versus Intermittent Boluses and Morphine Consumption: A Randomized, Blinded, Controlled Clinical Trial. Anesth Analg. 2018 Jun;126(6):2069-2077. doi: 10.1213/ANE.0000000000002747. PMID 29293181
- [Result] Jagannathan R, Niesen AD, D'Souza RS, Johnson RL. Intermittent bolus versus continuous infusion techniques for local anesthetic delivery in peripheral and truncal nerve analgesia: the current state of evidence. Reg Anesth Pain Med. 2019 Apr;44(4):447-451. doi: 10.1136/rapm-2018-100082. Epub 2019 Feb 3. PMID 30914472